CLINICAL TRIAL: NCT04622345
Title: A Single-Center, Double-Masked, Randomized, Placebo-Controlled, Phase 2, Evaluation of the Safety and Efficacy of VSJ-110 Ophthalmic Solution in the Treatment of Allergic Conjunctivitis Using an Allergen Challenge Model
Brief Title: Safety and Efficacy of VSJ-110 in the Treatment of Allergic Conjunctivitis in Adults With a History of Ocular Allergies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VP-VSJ-110-2101
Record Dates: First submitted 2020-11-04; First posted 2020-11-09 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2022-04

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VSJ-110 Solution (Experimental)
  Interventions: Drug: VSJ-110
- Placebo Solution (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VSJ-110 — ophthalmic solution
  Arms: VSJ-110 Solution
Drug: Placebo — ophthalmic solution
  Arms: Placebo Solution

SUMMARY:
The purpose of this study is to determine the safety and efficacy of VSJ-110 compared to placebo in the treatment of allergic conjunctivitis using an antigen challenge model

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age of either gender and any race
* Able to provide written informed consent and sign the HIPAA form
* Willing and able to follow all instructions and attend all study visits

Exclusion Criteria:

* Able and willing to avoid all disallowed medications during washout and study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-11-21 (Actual); Primary Completion 2021-05-22 (Actual); Study Completion 2021-06-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanda Investigational Site, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- VSJ-110: VSJ-110 Ophthalmic Solution
- Placebo: Placebo Ophthalmic Solution
Period: Overall Study
Arm/Group | VSJ-110 | Placebo
Started | 24 | 23
Completed | 22 | 18
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VSJ-110 | Placebo | Total
Number analyzed (Participants) | 24 | 23 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 21 | 40
  >=65 years | 5 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 9 | 11 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Number Analyzed: American Indian or Alaska Native | 0 | 1 | 1
  Number Analyzed: Asian | 0 | 0 | 0
  Number Analyzed: Black or African American | 0 | 2 | 2
  Number Analyzed: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Number Analyzed: White | 23 | 19 | 42
  Number Analyzed: Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching as Measured by Self-reported Numerical Scales
Description: Change from baseline in ocular itching evaluated by the subject at 3(±1), 5(±1), and 7(±1) minutes post allergen challenge (0-4 scale, with a higher number indicating more itching)
Time Frame: 16 hours, 8 hours, and 15 minutes post-treatment
Population: Efficacy analysis performed on ITT and PP populations
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | VSJ-110 | Placebo
Number analyzed (Participants) | 24 | 23
score on a scale
  16 hours (3(±1) minutes post-challenge) | -0.228 [-0.549 to 0.093] | 0.010 [-0.318 to 0.337]
  16 hours (5(±1) minutes post-challenge) | -0.424 [-0.731 to -0.118] | -0.035 [-0.349 to 0.278]
  16 hours (7(±1) minutes post-challenge) | -0.450 [-0.711 to -0.190] | -0.182 [-0.448 to 0.084]
  8 hours (3(±1) minutes post-challenge): number analyzed (Participants) | 23 | 21
  8 hours (3(±1) minutes post-challenge) | -0.383 [-0.762 to -0.004] | -0.402 [-0.799 to -0.006]
  8 hours (5(±1) minutes post-challenge): number analyzed (Participants) | 23 | 21
  8 hours (5(±1) minutes post-challenge) | -0.593 [-0.984 to -0.201] | -0.569 [-0.988 to -0.149]
  8 hours (7(±1) minutes post-challenge): number analyzed (Participants) | 23 | 21
  8 hours (7(±1) minutes post-challenge) | -0.698 [-1.073 to -0.322] | -0.772 [-1.165 to -0.379]
  15 minutes (3(±1) minutes post-challenge): number analyzed (Participants) | 23 | 20
  15 minutes (3(±1) minutes post-challenge) | 0.039 [-0.272 to 0.349] | -0.007 [-0.340 to 0.326]
  15 minutes (5(±1) minutes post-challenge): number analyzed (Participants) | 23 | 20
  15 minutes (5(±1) minutes post-challenge) | -0.248 [-0.588 to 0.093] | -0.140 [-0.505 to 0.225]
  15 minutes (7(±1) minutes post-challenge): number analyzed (Participants) | 23 | 20
  15 minutes (7(±1) minutes post-challenge) | -0.422 [-0.767 to -0.077] | -0.314 [-0.684 to 0.056]

2. Primary Outcome: Conjunctival Redness as Measured by Investigator Assessed Numerical Scales
Description: Change from baseline in conjunctival redness evaluated by the investigator at 7 (±1), 15 (±1), and 20 (±1) minutes post allergen challenge (0-4 scale, with a higher number indicating more redness)
Time Frame: 16 hours, 8 hours, and 15 minutes post-treatment
Population: Efficacy analysis performed on ITT and PP populations
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | VSJ-110 | Placebo
Number analyzed (Participants) | 24 | 23
score on a scale
  16 hours (7(±1) minutes post-challenge) | -0.280 [-0.523 to -0.036] | 0.075 [-0.174 to 0.323]
  16 hours (15(±1) minutes post-challenge) | -0.366 [-0.572 to -0.160] | -0.108 [-0.318 to 0.103]
  16 hours (20(±1) minutes post-challenge) | -0.491 [-0.713 to -0.268] | -0.151 [-0.379 to 0.076]
  8 hours (7(±1) minutes post-challenge): number analyzed (Participants) | 23 | 21
  8 hours (7(±1) minutes post-challenge) | -0.171 [-0.354 to 0.013] | -0.075 [-0.267 to 0.117]
  8 hours (15(±1) minutes post-challenge): number analyzed (Participants) | 23 | 21
  8 hours (15(±1) minutes post-challenge) | -0.208 [-0.359 to -0.057] | -0.201 [-0.359 to -0.043]
  8 hours (20(±1) minutes post-challenge): number analyzed (Participants) | 23 | 21
  8 hours (20(±1) minutes post-challenge) | -0.206 [-0.343 to -0.068] | -0.203 [-0.348 to -0.059]
  15 minutes (7(±1) minutes post-challenge): number analyzed (Participants) | 23 | 20
  15 minutes (7(±1) minutes post-challenge) | 0.162 [-0.011 to 0.334] | 0.252 [0.066 to 0.437]
  15 minutes (15(±1) minutes post-challenge): number analyzed (Participants) | 23 | 20
  15 minutes (15(±1) minutes post-challenge) | 0.039 [-0.157 to 0.236] | 0.030 [-0.181 to 0.241]
  15 minutes (20(±1) minutes post-challenge): number analyzed (Participants) | 23 | 20
  15 minutes (20(±1) minutes post-challenge) | 0.002 [-0.180 to 0.185] | 0.035 [-0.161 to 0.231]

3. Secondary Outcome: Conjunctival Redness Responder Rates as Evaluated by the Investigator Using Numerical Scales
Description: Conjunctival redness responder rates evaluated by the investigator at 7(±1), 15(±1), and 20(±1) minutes post allergen challenge. A responder is defined as meeting 1, 1.5, or 2 points reduction from baseline, or complete response in all three time points or at least two out of the three timepoints.
Time Frame: 16 hours, 8 hours, and 15 minutes post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | VSJ-110 | Placebo
Number analyzed (Participants) | 24 | 23
Participants
  16 hours (rates across all three time points) | 3 | 0
  8 hours (rates across all three time points) | 1 | 0
  15 minutes (rates across all three time points) | 0 | 0
  16 hours (rates across two out of the three timepoints) | 5 | 1
  8 hours (rates across two out of the three timepoints) | 1 | 0
  15 minutes (rates across two out of the three timepoints) | 0 | 1

ADVERSE EVENTS:
Time Frame: AE data was collected during the 4 week treatment period plus a 7 day follow up period.
Arm/Group | VSJ-110 Solution | Placebo Solution
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/24 | 1/23
Other Adverse Events (participants affected / at risk) | 2/24 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VSJ-110 Solution (N=24) | Placebo Solution (N=23)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VSJ-110 Solution (N=24) | Placebo Solution (N=23)
Visual acuity reduced (Eye disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT04622345/Prot_SAP_000.pdf